CLINICAL TRIAL: NCT02606461
Title: A Phase 2-3, Multicenter, Randomized, Double-blind Study of Selinexor (KPT-330) Versus Placebo in Patients With Advanced Unresectable Dedifferentiated Liposarcoma (DDLS)
Brief Title: Selinexor in Advanced Liposarcoma
Acronym: SEAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KCP-330-020; 2015-003594-14 (EudraCT Number)
Record Dates: First submitted 2015-10-13; First posted 2015-11-17 (Estimated); Results first posted 2021-12-07 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Dedifferentiated Liposarcoma
Keywords: Advanced unresectable dedifferentiated liposarcoma; selinexor; KCP-330; Karyopharm; Phase 2 / 3; dedifferentiated liposarcoma; Liposarcoma
MeSH Terms: conditions — Liposarcoma | interventions — selinexor; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 2 Double-blinded: Selinexor (Experimental): Participants received a fixed blinding dose of 60 milligrams (mg) selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle until progressive disease (PD).
  Interventions: Drug: Selinexor
- Phase 3 Double-blinded: Selinexor (Experimental): Participants received a fixed blinding dose of 60 mg selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle until PD.
  Interventions: Drug: Selinexor
- Phase 2 Double-blinded: Placebo Followed by Open Label- Selinexor (Placebo Comparator): Participants received a fixed blinding dose of placebo matched to selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle until PD in double-blinded treatment period. Participants in the placebo group who had PD during the Phase 2 double-blinded treatment, will be elected to cross over to open-label selinexor.
  Interventions: Drug: Placebo
- Phase 3 Double-blinded: Placebo Followed by Open Label- Selinexor (Placebo Comparator): Participants received a fixed blinding dose of placebo matched to selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle until PD or development of unacceptable toxicity. Participants in the placebo group who had PD during the Phase 3 double-blinded treatment, will be elected to cross over to open-label selinexor.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selinexor — Selinexor 60mg
  Other Names: KPT-330
  Arms: Phase 2 Double-blinded: Selinexor; Phase 3 Double-blinded: Selinexor
Drug: Placebo
  Other Names: sugar pill
  Arms: Phase 2 Double-blinded: Placebo Followed by Open Label- Selinexor; Phase 3 Double-blinded: Placebo Followed by Open Label- Selinexor

SUMMARY:
This is a randomized, multicenter, double-blind, placebo-controlled, Phase 2-3 study of patients diagnosed with advanced unresectable dedifferentiated liposarcoma. Approximately 342 total patients will be randomized to study treatment (selinexor or placebo).

DETAILED DESCRIPTION:
In the Phase 2 portion of the study, 57 patients were randomized to selinexor (60 mg) or placebo at a 1:1 allocation ratio.

In the Phase 3 portion of the study, approximately 285 patients will be randomized to selinexor (60 mg) or placebo with a 2:1 allocation ratio.

Patients who progress during the blinded portion of the study will be unblinded and if receiving:

* placebo, may cross over to open-label selinexor (60mg twice-weekly)
* selinexor, will be withdrawn from further treatment and followed for survival

Study treatment will be given twice-weekly on Day 1 and Day 3 during Weeks 1-6 of each six-week (42 day) cycle until disease progression or intolerability.

Treatment will continue until one or more of the following occurs:

* Disease progression, as defined by RECIST v1.1 Response Criteria
* Clinical progression, as determined by the treating physician
* Unacceptable adverse events (AEs) or failure to tolerate study treatment
* Patient withdrawal
* Patient discontinuation due to non-compliance

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥12 years of age
2. Body surface area (BSA) ≥ 1.2 m2
3. Histologic evidence of DDLS at any time prior to randomization AND current evidence of DDLS requiring treatment
4. Must have measurable disease per RECIST v1.1 Response Criteria
5. Radiologic evidence of disease progression within 6 months prior to randomization. If the patient received other intervening therapy after documented disease progression, further disease progression must be documented after the completion of the intervening therapy
6. Must have had at least 2 prior lines of systemic therapy for liposarcoma (not to exceed 5 prior lines)
7. If patient received any previous systemic therapy, the last dose must have been ≥ 21 days prior to randomization (or ≥ 5 half-lives of that drug, whichever is shorter) with all clinically significant therapy-related toxicities having resolved to ≤ Grade 1

Exclusion Criteria:

1. Patients with pure well-differentiated liposarcoma (WDLS), myxoid/round cell or pleomorphic tumor histologic subtypes
2. Known active hepatitis B (HepB), hepatitis C (HepC) or human immunodeficiency virus (HIV) infection
3. Known central nervous system metastases

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (26):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford University, Stanford, California
  - University of Colorado-Denver, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Northwell Health Physicians Partners, New York, New York
  - Duke Institute of Cancer, Durham, North Carolina
  - James Cancer Center, Ohio State University, Columbus, Ohio
  - Oregon Health and Science, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Vanderbilt, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (3):
  - UZ Brussel, Brussels
  - UCL Saint-Luc, Brussels
  - UZ Gent, Ghent
- Canada (4):
  - Cross Cancer Center - Alberta Health Services, Edmonton, Alberta
  - The Ottawa Hospital Cancer, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- France (9):
  - Institut Bergonie, Bordeaux
  - Oscar Lambret Center, Lille
  - Centre Leon Berard, Lyon
  - Timone University Hospital, Marseille
  - Institut Régional du Cancer de Montpellier (ICM), Montpellier
  - CLCC Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Helios Hospital Berlin-Buch, Berlin
  - Technische Universitaet Dresden Med. Fakultaet Carl Gustav Carus Med. Klinik u. Poliklinik I, Dresden
  - National Center for Tumor Diseases, Univeristy Hospital Heidelberg, Heidelberg
  - University Hospital Mannheim, Mannheim
  - Klinik und Poliklinik für Innere Medizin III, Hämatologie und Onkologie Klinikum rechts der Isar der TU Muenchen, München
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical, Tel Aviv
  - Assaf Harofe Medical Center, Ẕerifin
- Italy (4):
  - Candiolo Cancer Institute, Candiolo
  - Istituto Nazionale dei Tumori, Milan, Milan
  - U.O.C. Oncologia Medica Oncology Department, Palermo
  - Policlinico Universitario Campus Biomedico, Roma
- Spain (7):
  - "Germans Trias Pujol" University Hospital, Badalona
  - Vall d´hebron University Hospital, Barcelona
  - Hospital Sant Pau Barcelona, Barcelona
  - Hospital ICO Bellvitge, Barcelona
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital La Fe Valencia, Valencia
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skane University Hospital, Lund
  - Onkologiska Kliniken, Stockholm
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University College London Hospitals, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gounder MM, Razak AA, Somaiah N, Chawla S, Martin-Broto J, Grignani G, Schuetze SM, Vincenzi B, Wagner AJ, Chmielowski B, Jones RL, Riedel RF, Stacchiotti S, Loggers ET, Ganjoo KN, Le Cesne A, Italiano A, Garcia Del Muro X, Burgess M, Piperno-Neumann S, Ryan C, Mulcahy MF, Forscher C, Penel N, Okuno S, Elias A, Hartner L, Philip T, Alcindor T, Kasper B, Reichardt P, Lapeire L, Blay JY, Chevreau C, Valverde Morales CM, Schwartz GK, Chen JL, Deshpande H, Davis EJ, Nicholas G, Groschel S, Hatcher H, Duffaud F, Herraez AC, Beveridge RD, Badalamenti G, Eriksson M, Meyer C, von Mehren M, Van Tine BA, Gotze K, Mazzeo F, Yakobson A, Zick A, Lee A, Gonzalez AE, Napolitano A, Dickson MA, Michel D, Meng C, Li L, Liu J, Ben-Shahar O, Van Domelen DR, Walker CJ, Chang H, Landesman Y, Shah JJ, Shacham S, Kauffman MG, Attia S. Selinexor in Advanced, Metastatic Dedifferentiated Liposarcoma: A Multinational, Randomized, Double-Blind, Placebo-Controlled Trial. J Clin Oncol. 2022 Aug 1;40(22):2479-2490. doi: 10.1200/JCO.21.01829. Epub 2022 Apr 8. PMID 35394800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 71 sites in the United States, Canada, Germany, Belgium, Israel, United Kingdom, France, Spain, Italy, and Sweden. A total of 342 participants were enrolled, out of which 57 participants were randomized to receive study treatment in Phase 2 and 285 participants randomized, of which 284 participants received study treatment in Phase 3.
Pre-assignment Details: This study consisted of 2 phases (2 and 3), where participants were randomized to selinexor or placebo in double-blind treatment. Participants in the placebo group who had progressive disease (PD) during the phase 2 and 3 double-blinded treatment could crossover to open-label selinexor treatment.
Groups:
- Phase 2 Double-blinded: Selinexor: Participants received a fixed blinding dose of 60 milligrams (mg) selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle.
- Phase 2 Double-blinded: Placebo; Phase 3 Double-blinded: Placebo: Participants received a fixed blinding dose of placebo matched to selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle.
- Phase 3 Double-blinded: Selinexor: Participants received a fixed blinding dose of 60 mg selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle.
- Phase 2 Open-label: Selinexor: Participants in the placebo group who had PD during Phase 2 double-blinded treatment were entered in open-label and received selinexor 60 mg tablet twice-weekly during Weeks 1 to 6 of each 6-week (42-day) cycle.
- Phase 3 Open-label: Selinexor: Participants in the placebo group who had PD during Phase 3 double-blinded treatment, were entered in open-label and received selinexor 60 mg tablet twice-weekly during Weeks 1 to 6 of each 6-week (42-day) cycle.
Period: Period 1: Double-blinded Period
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo | Phase 2 Open-label: Selinexor | Phase 3 Open-label: Selinexor
Started | 27 | 30 | 188 | 97 | 0 | 0
Treated | 27 | 30 | 187 | 97 | 0 | 0
Completed | 27 | 30 | 187 | 97 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Randomized but no treatment | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2: Open Label Period
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo | Phase 2 Open-label: Selinexor | Phase 3 Open-label: Selinexor
Started | 0 | 0 | 0 | 0 | 24 (Participants in the placebo group who had PD during the Phase 2 double-blinded treatment, switched to open-label selinexor.) | 63 (Participants in the placebo group who had PD during the Phase 3 double-blinded treatment, switched to open-label selinexor.)
Completed | 0 | 0 | 0 | 0 | 24 | 63
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 Double-blinded: Selinexor; Phase 3 Double-blinded: Selinexor: Participants received a fixed blinding dose of 60 mg selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo | Total
Number analyzed (Participants) | 27 | 30 | 188 | 97 | 342
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 17 | 92 | 46 | 174
  >=65 years | 8 | 13 | 96 | 51 | 168
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 74 | 33 | 130
  Male | 15 | 19 | 114 | 64 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 7 | 6 | 18
  Not Hispanic or Latino | 25 | 25 | 149 | 79 | 278
  Unknown or Not Reported | 0 | 2 | 32 | 12 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 5 | 9 | 3 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 0 | 3
  Black or African American | 1 | 2 | 3 | 1 | 7
  White | 23 | 20 | 139 | 80 | 262
  More than one race | 0 | 3 | 34 | 13 | 50
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 3 Double Blind: Progression-free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS was defined as the time from the date of randomization until the first date of Independent Review Committee (IRC)-confirmed PD per RECIST version 1.1, or death due to any cause. PD was defined as at least a 20% increase in the sum of the longest diameter (SLD), taking as reference the smallest sum of the longest diameter (SLD) recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization until the first date of disease progression, or death due to any cause whichever occurred first (up to 57 months)
Population: Phase 3 Intent-to-Treat Population (Ph3-ITT) consisted of all participants randomized to study treatment in Phase 3, regardless of whether or not they received study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 188 | 97
Months | 2.83 [2.73 to 4.11] | 2.07 [1.51 to 3.06]
Statistical Analysis 1: Comparison: Phase 3 Double-blinded: Selinexor vs Phase 3 Double-blinded: Placebo; Test type: Superiority; p = 0.0114, Log Rank; Hazard Ratio (HR) = 0.7026, 95% CI 2-sided [0.5191 to 0.9509]

2. Primary Outcome: Phase 3 Open Label: Progression-free Survival (PFS) as Per RECIST Version 1.1
Description: PFS was defined as the time from the date of randomization in the Phase 3 open-label period until the first date of IRC-confirmed PD per RECIST version 1.1, or death due to any cause. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization in the Phase 3 open label period until the first date of disease progression, or death due to any cause whichever occurred first (up to 57 months)
Population: The Phase 3 Open-Label Population (Ph3-OL) consisted of all participants in Phase 3 who were randomized to placebo in the blinded phase, entered the open-label period, and received at least one dose of open-label selinexor.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 3 Open Label: Selinexor: Participants in the placebo group who had PD during Phase 3 double-blinded treatment, were entered in open-label and received selinexor 60 mg tablet twice-weekly during Weeks 1 to 6 of each 6-week (42-day) cycle.
Arm/Group | Phase 3 Open Label: Selinexor
Number analyzed (Participants) | 63
Months | 2.73 [1.97 to 4.14]

3. Primary Outcome: Phase 2 Double Blind: Progression-free Survival (PFS) as Per RECIST Version 1.1
Description: PFS was defined as the time from date of randomization until the first date of IRC-confirmed PD per RECIST version 1.1, or death due to any cause. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From date of randomization until the first date of PD or death due to any cause, whichever occurred first (up to 57 months)
Population: The Phase 2 Intent-to-Treat Population (Ph2-ITT) consisted of all participants randomized to study treatment in Phase 2, regardless of whether or not they received study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo
Number analyzed (Participants) | 27 | 30
Months | 3.02 [1.41 to NA] — Data could not be estimated due to higher number (>50%) of deaths. | 2.76 [1.58 to NA] — Data could not be estimated due to higher number (>50%) of deaths.
Statistical Analysis 1: Comparison: Phase 2 Double-blinded: Selinexor vs Phase 2 Double-blinded: Placebo; Test type: Superiority; p = 0.6051, Log Rank; Hazard Ratio, log = 1.1521, 95% CI 2-sided [0.5357 to 2.4778]

4. Primary Outcome: Phase 2 Open Label: Progression-free Survival (PFS) as Per RECIST Version 1.1
Description: PFS was defined as the time from date of randomization in the Phase 2 open-label period until the first date of IRC-confirmed PD per RECIST version 1.1, or death due to any cause. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From date of randomization in the Phase 2 open label period until the first date of PD or death due to any cause, whichever occurred first (up to 57 months)
Population: The Phase 2 Open-Label Population (Ph2-OL) consisted of all participants in Phase 2 who were randomized to placebo in the blinded phase, entered open-label period, and received at least one dose of open-label selinexor.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 2 Open Label: Selinexor: Participants in the placebo group who had PD during Phase 2 double-blinded treatment were entered in open-label and received selinexor 60 mg tablet twice-weekly during Weeks 1 to 6 of each 6-week (42-day) cycle.
Arm/Group | Phase 2 Open Label: Selinexor
Number analyzed (Participants) | 24
Months | 1.38 [1.38 to 2.27]

5. Secondary Outcome: Phase 3 Double Blind: Overall Survival (OS)
Description: OS was defined as the duration (in months) from the date of randomization to death from any cause. Participants last known to be alive were censored at the date of discontinuation from the study, or database cut date, whichever was earlier.
Time Frame: From date of randomization until death due to any cause, whichever occurred first (up to 70 months)
Population: The Ph3-ITT consisted of all participants randomized to study treatment in Phase 3, regardless of whether or not they received study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 188 | 97
Months | 10.38 [8.41 to 13.40] | 12.71 [8.54 to 15.90]

6. Secondary Outcome: Phase 3 Open Label: Overall Survival (OS)
Description: OS was defined as the duration (in months) from the date of randomization in the Phase 3 open-label period to death from any cause. Participants last known to be alive were censored at the date of discontinuation from the study, or database cut date, whichever was earlier.
Time Frame: From date of randomization in phase 3 open label period until death due to any cause, whichever occurred first (up to 70 months)
Population: The Ph3-OL consisted of all participants in Phase 3 who were randomized to placebo in the blinded phase, entered the open-label period, and received at least one dose of open-label selinexor.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3 Open Label: Selinexor
Number analyzed (Participants) | 63
Months | 10.18 [5.78 to 14.69]

7. Secondary Outcome: Phase 2 Double Blind: Overall Survival (OS)
Description: as for outcome 5
Time Frame: From the date of randomization until death due to any cause, whichever occurred first (up to 70 months)
Population: The Ph2-ITT consisted of all participants randomized to study treatment in Phase 2, regardless of whether or not they received study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 2 Double-blinded: Placebo: Participants received a fixed blinding dose of 60 mg selinexor twice-weekly on Day 1 and 3 during each 6-week (42-day) cycle.
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo
Number analyzed (Participants) | 27 | 30
Months | 17.31 [10.51 to 29.57] | 16.07 [8.38 to 23.06]

8. Secondary Outcome: Phase 2 Open Label: Overall Survival (OS)
Description: OS was defined as the duration (in months) from the date of randomization in the Phase 2 open-label period to death from any cause. Participants last known to be alive were censored at the date of discontinuation from the study, or database cut date, whichever was earlier.
Time Frame: From date of randomization in the Phase 2 open-label period until death due to any cause, whichever occurred first (up to 70 months)
Population: The Ph2-OL consisted of all participants in Phase 2 who were randomized to placebo in the blinded phase, entered the open-label period, and received at least one dose of open-label selinexor.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Open Label: Selinexor
Number analyzed (Participants) | 24
Months | 8.90 [4.96 to 18.92]

9. Secondary Outcome: Phase 3 Double Blind: Time-to-Progression (TTP) as Per RECIST Version 1.1
Description: TTP was defined as the time from date of randomization until ICR-determined PD per RECIST version 1.1, or death due to disease progression, whichever occurred first. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From date of randomization until the first date of PD or death due to any cause, whichever occurred first (up to 70 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 188 | 97
Months | 2.83 [2.73 to 4.11] | 2.10 [1.51 to 3.06]

10. Secondary Outcome: Phase 3 Open Label: Time-to-Progression (TTP) as Per RECIST Version 1.1
Description: TTP was defined as the time from date of randomization in the Phase 3 open-label period until ICR-determined PD per RECIST version 1.1, or death due to disease progression, whichever occurred first. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From date of randomization in the Phase 3 open label period until the first date of PD or death due to any cause, whichever occurred first (up to 70 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3 Open Label: Selinexor
Number analyzed (Participants) | 63
Months | 2.73 [1.97 to 4.14]

11. Secondary Outcome: Phase 2 Double Blind: Time-to-Progression (TTP) as Per RECIST Version 1.1
Description: TTP was defined as the time from date of randomization until ICR-determined PD as per RECIST version 1.1, or death due to disease progression, whichever occurred first. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: as for outcome 9
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo
Number analyzed (Participants) | 27 | 30
Months | 3.02 [1.41 to NA] — Data could not be estimated due to the higher number (>50%) of deaths. | 2.76 [1.58 to NA] — Data could not be estimated due to the higher number (>50%) of deaths.

12. Secondary Outcome: Phase 2 Open Label: Time-to-Progression (TTP) as Per RECIST Version 1.1
Description: TTP was defined as the time from date of randomization in the Phase 2 open-label period until ICR-determined PD per RECIST version 1.1, or death due to disease progression, whichever occurred first. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From date of randomization in the Phase 2 open-label period until the first date of PD or death due to any cause, whichever occurred first (up to 70 months)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Open Label: Selinexor
Number analyzed (Participants) | 24
Months | 1.38 [1.38 to 2.27]

13. Secondary Outcome: Phase 3 Double Blind: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved complete response (CR) or partial response (PR), per RECIST v.1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization until the documentation of CR or PR (up to 70 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 188 | 97
Percentage of participants | 2.7 [0.9 to 6.1] | 0 [NA to NA] — Data could not be evaluated due to no CR or PR events in the placebo arm.

14. Secondary Outcome: Phase 3 Open Label: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved CR or PR, per RECIST v.1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization in the Phase 3 open label period until the documentation of CR or PR (up to 70 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3 Open Label: Selinexor
Number analyzed (Participants) | 63
Percentage of participants | 3.2 [0.4 to 11]

15. Secondary Outcome: Phase 2 Double Blind: Overall Response Rate (ORR)
Description: as for outcome 14
Time Frame: From date of randomization until the documentation of CR or PR (up to 70 months)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo
Number analyzed (Participants) | 27 | 30
Percentage of participants | 0 [NA to NA] — Data could not be evaluated since no participant had CR or PR. | 0 [NA to NA] — Data could not be evaluated since no participant had CR or PR.

16. Secondary Outcome: Phase 2 Open Label: Overall Response Rate (ORR)
Description: as for outcome 14
Time Frame: From date of randomization in the Phase 2 open-label period until the documentation of CR or PR (up to 70 months)
Population: The Ph2-OL consisted of all participants in Phase 2 who were randomized to placebo in the blinded phase, entered the open-label period, and received at least one dose of open-label selinexor. Data could not be evaluated due to no CR or PR events.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 2 Open Label: Selinexor
Number analyzed (Participants) | 24
Percentage of participants
  Participants who achieved CR | 0
  Participants who achieved PR | 0

17. Secondary Outcome: Phase 3 Double Blind: Duration of Response (DOR)
Description: DOR was defined as the time from first occurrence of CR or PR until the first date of PD per RECIST version 1.1 or death. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From first occurrence of CR or PR until the first date of PD (up to 70 months)
Population: The Ph3-ITT consisted of all participants randomized to study treatment in Phase 3, regardless of whether or not they received study treatment. Here, "overall number of participants analyzed" signifies those who had CR and PR in specified group/arm and phase.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 5 | 0
Months | 7.39 [NA to NA] — Upper and lower limit of 95% CI was not estimable due to lesser number of participants with events. |

18. Secondary Outcome: Phase 3 Double Blind: Progression-free Survival (PFS) as Per Investigator Assessment
Description: PFS was defined as the time from date of randomization until the first date of PD, per RECIST version 1.1, or death due to any cause as defined by the Investigator based on clinical and/or radiologic criteria. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization until the first date of disease progression, or death due to any cause whichever occurred first (up to 70 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 188 | 97
Months | 2.89 [2.76 to 4.17] | 1.87 [1.45 to 2.89]

19. Secondary Outcome: Phase 3 Double Blind: Time to Next Treatment (TTNT)
Description: TTNT was defined as time since randomization until the first new antineoplastic therapy or death due to any cause, whichever occurs first.
Time Frame: Time from randomization to the first new antineoplastic therapy or death due to any cause (up to 70 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 188 | 97
Months | 5.42 [4.67 to 6.34] | 3.22 [2.56 to 3.78]

20. Secondary Outcome: Phase 2 Double Blind: Time to Next Treatment (TTNT)
Description: as for outcome 19
Time Frame: Time from randomization to the first new antineoplastic therapy or death due to any cause (up to 70 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo
Number analyzed (Participants) | 27 | 30
Months | 4.96 [3.91 to 14.03] | 2.92 [2.04 to 5.06]

21. Secondary Outcome: Phase 3 Double Blind: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. A TEAE was defined as those AEs that develop or worsen after the first dose of study drug. TEAEs included both serious and non-serious TEAEs.
Time Frame: From start of study drug administration up to 70 months
Population: The Phase 3 Safety Population (Ph3-SAF) consisted of all participants in Phase 3 who had received at least one dose of blinded study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 187 | 97
Participants
  Participants with TEAEs | 187 | 94
  Participants with Serious TEAEs | 73 | 18

22. Secondary Outcome: Phase 3 Open Label: Number of Participants With TEAEs and Serious TEAEs
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as those AEs that develop or worsen after the first dose of study drug. TEAEs included both serious and non-serious TEAEs.
Time Frame: From start of study drug administration up to 70 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3 Open Label: Selinexor
Number analyzed (Participants) | 63
Participants
  Participants with TEAEs | 63
  Participants with Serious TEAEs | 25

23. Secondary Outcome: Phase 2 Double Blind: Number of Participants With TEAEs and Serious TEAEs
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as those AEs that develop or worsen after the first dose of study drug. TEAEs included both serious and non-serious TEAEs.
Time Frame: From start of study drug administration up to 70 months
Population: The Phase 2 Safety Population (Ph2-SAF) consisted of all participants in Phase 2 who had received at least one dose of blinded study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo
Number analyzed (Participants) | 27 | 30
Participants
  Participants with TEAEs | 27 | 29
  Participants with Serious TEAEs | 4 | 6

24. Secondary Outcome: Phase 2 Open Label: Number of Participants With TEAEs and Serious TEAEs
Description: as for outcome 22
Time Frame: From start of study drug administration up to 70 months
Population: The Ph2-OL consisted of all participants in Phase 2 who were randomized to placebo in the blinded phase, entered open-label period, and received at least one dose of open-label selinexor.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Open Label: Selinexor
Number analyzed (Participants) | 24
Participants
  Participants with TEAEs | 24
  Participants with Serious TEAEs | 13

25. Secondary Outcome: Phase 3 Double Blind: Change From Baseline in Quality-of-life Questionnaire 30 Item (QLQ-C30)
Description: The QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of patients with cancer. QLQ-C30 contains 30 questions that include five functional scales (physical, role, emotional, social, and cognitive functioning); three symptom scales (fatigue, nausea/vomiting and pain); six single-item symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties); and global health status/quality of life (QoL). Most questions used a 4-point scale (from 1 'Not at all' to 4 'Very much'); 2 questions used a 7-point scale (from 1 'very poor' to 7 'Excellent'). Scores were averaged and transformed to a 0-100 scale. For the functional scales and the global health status/QoL, a higher score represents a better level of functioning (better health status); for the symptom scales/items, a higher score represents a higher level of symptomatology/problems (worse health status).
Time Frame: Baseline up to Day 1387
Population: The Ph3-ITT consisted of all participants randomized to study treatment in Phase 3, regardless of whether or not they received study treatment. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo
Number analyzed (Participants) | 1 | 0
Score on a Scale
  Global Health Status | 33.33 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Physical Functioning | 20.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Role Functioning | 16.67 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Emotional Functioning | 8.33 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Social Functioning | 50.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Cognitive Functioning | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Fatigue | -22.22 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Nausea and Vomiting | 16.67 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Pain | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Dyspnoea | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Insomnia | 33.33 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Appetite Loss | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Constipation | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Diarrhoea | 33.33 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |
  Financial Difficulties | -66.67 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant. |

26. Secondary Outcome: Phase 3 Open Label: Change From Baseline in Quality-of-life Questionnaire 30 Item (QLQ-C30)
Description: as for outcome 25
Time Frame: Baseline up to Day 379
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Phase 3 Open Label: Selinexor
Number analyzed (Participants) | 1
Score on a Scale
  Global Health Status | -16.67 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Physical Functioning | -40.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Role Functioning | -33.33 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Emotional Functioning | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Social Functioning | -50.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Cognitive Functioning | -16.67 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Fatigue | 66.67 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Nausea and Vomiting | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Pain | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Dyspnoea | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Insomnia | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Appetite Loss | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Constipation | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Diarrhoea | 0.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.
  Financial Difficulties | 100.00 (NA) — Here, "NA" signifies standard deviation was not estimated due to single participant.

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 70 months
Description: The Ph2-SAF and Ph3-SA consisted of all participants who had received at least one dose of blinded study treatment in Phase 2 and Phase 3 respectively. The Phase 3 open-label population (Ph3-OL) and Phase 2 open-label Population (Ph2-OL) consisted of all participants in Phase 3 and Phase 2 respectively, who were randomized to placebo in the blinded phase, entered the open-label period, and received at least one dose of open-label selinexor.
Arm/Group | Phase 2 Double-blinded: Selinexor | Phase 2 Double-blinded: Placebo | Phase 3 Double-blinded: Selinexor | Phase 3 Double-blinded: Placebo | Phase 2 Open-label: Selinexor | Phase 3 Open-label: Selinexor
All-Cause Mortality (participants affected / at risk) | 18/27 | 25/30 | 127/187 | 67/97 | 20/24 | 43/63
Serious Adverse Events (participants affected / at risk) | 4/27 | 6/30 | 73/187 | 18/97 | 13/24 | 25/63
Other Adverse Events (participants affected / at risk) | 27/27 | 29/30 | 186/187 | 94/97 | 24/24 | 62/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2 Double-blinded: Selinexor (N=27) | Phase 2 Double-blinded: Placebo (N=30) | Phase 3 Double-blinded: Selinexor (N=187) | Phase 3 Double-blinded: Placebo (N=97) | Phase 2 Open-label: Selinexor (N=24) | Phase 3 Open-label: Selinexor (N=63)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 1 | 2 | 0 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Small intestine obstruction (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 7 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Anastomotic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 3 | 0 | 2 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 3 | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2 Double-blinded: Selinexor (N=27) | Phase 2 Double-blinded: Placebo (N=30) | Phase 3 Double-blinded: Selinexor (N=187) | Phase 3 Double-blinded: Placebo (N=97) | Phase 2 Open-label: Selinexor (N=24) | Phase 3 Open-label: Selinexor (N=63)
Anaemia (Blood and lymphatic system disorders) | 16 | 9 | 91 | 22 | 10 | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 2 | 72 | 5 | 11 | 24
Leukopenia (Blood and lymphatic system disorders) | 9 | 1 | 26 | 1 | 5 | 13
Neutropenia (Blood and lymphatic system disorders) | 8 | 1 | 38 | 1 | 6 | 12
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 14 | 4 | 1 | 6
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 7 | 6 | 1 | 6
Tachycardia (Cardiac disorders) | 2 | 0 | 3 | 3 | 0 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 4 | 2 | 2 | 0
Vision Blurred (Eye disorders) | 8 | 2 | 42 | 3 | 9 | 8
Cataract (Eye disorders) | 2 | 1 | 7 | 1 | 1 | 2
Photopsia (Eye disorders) | 2 | 0 | 9 | 0 | 1 | 1
Visual Impairement (Eye disorders) | 0 | 0 | 10 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 24 | 10 | 151 | 38 | 20 | 45
Vomiting (Gastrointestinal disorders) | 15 | 4 | 93 | 12 | 14 | 31
Abdominal pain (Gastrointestinal disorders) | 6 | 8 | 49 | 30 | 5 | 13
Constipation (Gastrointestinal disorders) | 6 | 8 | 74 | 23 | 6 | 14
Diarrhoea (Gastrointestinal disorders) | 8 | 5 | 75 | 17 | 7 | 18
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 11 | 6 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 10 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 11 | 1 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 18 | 6 | 1 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 11 | 1 | 1 | 0
Fatigue (General disorders) | 15 | 14 | 96 | 31 | 18 | 33
Oedema peripheral (General disorders) | 3 | 3 | 30 | 12 | 3 | 10
Pyrexia (General disorders) | 1 | 4 | 20 | 9 | 1 | 8
Influenza like illness (General disorders) | 1 | 3 | 3 | 1 | 1 | 0
Malaise (General disorders) | 3 | 1 | 2 | 2 | 3 | 1
Chills (General disorders) | 0 | 0 | 11 | 7 | 2 | 1
Pain (General disorders) | 1 | 2 | 4 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 5 | 2 | 1 | 2
Asthenia (General disorders) | 1 | 0 | 58 | 10 | 1 | 13
General physical health deterioration (General disorders) | 0 | 0 | 2 | 2 | 0 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 3 | 2 | 0 | 4
Urinary tract infection (Infections and infestations) | 5 | 3 | 13 | 8 | 3 | 4
Rhinitis (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 2 | 2 | 2
Weight decreased (Investigations) | 14 | 0 | 81 | 9 | 15 | 25
Blood alkaline phosphatase increased (Investigations) | 6 | 7 | 14 | 10 | 3 | 5
Alanine aminotransferase increased (Investigations) | 6 | 2 | 16 | 5 | 3 | 6
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 11 | 5 | 2 | 7
Activated partial thromboplastin time prolonged (Investigations) | 0 | 4 | 4 | 3 | 2 | 4
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 5 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 2 | 5 | 2 | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 15 | 5 | 144 | 21 | 14 | 32
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 6 | 52 | 8 | 10 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 3 | 21 | 8 | 2 | 7
Hypercreatininaemia (Metabolism and nutrition disorders) | 4 | 5 | 42 | 13 | 7 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 5 | 10 | 8 | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4 | 20 | 5 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 3 | 24 | 2 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0 | 8 | 4 | 1 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 13 | 2 | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 11 | 3 | 3 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 3 | 0 | 6 | 2 | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 13 | 3 | 1 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 2 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 26 | 12 | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 9 | 5 | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 11 | 2 | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 9 | 7 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 12 | 3 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 11 | 4 | 1 | 5
Dysgeusia (Nervous system disorders) | 10 | 2 | 51 | 4 | 6 | 12
Dizziness (Nervous system disorders) | 7 | 3 | 45 | 6 | 4 | 11
Headache (Nervous system disorders) | 4 | 3 | 23 | 3 | 3 | 7
Taste disorder (Nervous system disorders) | 3 | 0 | 8 | 1 | 2 | 5
Sciatica (Nervous system disorders) | 2 | 0 | 1 | 3 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 11 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 1 | 21 | 4 | 2 | 2
Anxiety (Psychiatric disorders) | 0 | 2 | 6 | 0 | 1 | 4
Depression (Psychiatric disorders) | 0 | 1 | 11 | 2 | 2 | 5
Confusional state (Psychiatric disorders) | 1 | 0 | 6 | 1 | 2 | 1
Haematuria (Renal and urinary disorders) | 3 | 0 | 7 | 7 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 2 | 0 | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 6 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 30 | 7 | 7 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 6 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 7 | 0 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 6 | 1 | 7 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 13 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 5 | 2 | 0
Hypertension (Vascular disorders) | 5 | 3 | 22 | 10 | 3 | 6
Hypotension (Vascular disorders) | 4 | 3 | 23 | 3 | 3 | 5
Hot flush (Vascular disorders) | 0 | 0 | 3 | 3 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT02606461/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT02606461/SAP_001.pdf